CLINICAL TRIAL: NCT01236157
Title: Monitoring of Nontraumatic Chest Pain Borne by the "Department of Emergency Help Medicalized" (SAMU)
Acronym: DOLORES
Status: Completed | Type: Observational
Sponsor: French Cardiology Society (Other)
Responsible Party: Principal Investigator, Spaulding Christian, Professor, French Cardiology Society
Other Study IDs: 09365
Record Dates: First submitted 2010-06-01; First posted 2010-11-08 (Estimated); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Chest Pain
Keywords: Cardiology
MeSH Terms: conditions — Chest Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Chest Pain: All patients that call to the SAMU-ACS because of chest pain are included

SUMMARY:
Support pre-hospital chest pain remains a difficult problem in both pre hospital regulation that when supported by the Mobile Services Emergency and Intensive Care (SMUR).

This ground of appeal underlying various pathologies especially acute coronary syndrome whose early care diagnostic and treatment significantly improves the prognosis.

The recognition and management of SCA is therefore a public health issue. Myocardial infarction (MI) is responsible for 10 to 12% of the total annual mortality in adults and coronary heart disease is the leading cause of death in France.

No studies have assessed the adequacy of regulation and management of chest pain SAMU for the diagnosis of SCA.

The main objective of the research is to have a descriptive analysis of the population controlled by the SAMU and the population served by the mobile emergency with chest pain. Also evaluate the adequacy of the proposed direction by the ambulance SAMU/SMUR and the final diagnosis and direction after passing emergency, cardiology and at follow-up to a year.

DETAILED DESCRIPTION:
Course of study:

* Call the ambulance dispatch center: anamnestic data will be collected by the regulator on a medical report forms The patient is identified by an anonymous number, "number of SAMU business". The CRA of Centre concerned, from this number of case (using the database of SAMU) capture, in the database of the French Society of Cardiology - FSC - the patient identification data (name , surname, date of birth, address, telephone number and the name and address of attending physician, these data will be necessary for the CRA to the FSC to follow up to 1 year)
* SMUR: if the patient arrives at SMUR, anamnestic data, clinical, laboratory, ECG, therapeutic, diagnostic and referral will be collected by the contact center on a paper CRF or on the computerized database of CFS by centers.
* Emergency Service: If the patient comes to the ER, the clinical, laboratory, ECG, diagnostic output will be collected on a paper CRF or the computerized database of CFS according to the center by the referent of Centre concerned.
* Cardiology service : if the patient arrives in the cardiology service, laboratory, ECG, diagnostic output will be collected on a paper CRF or the computerized database of CFS according to the center by the referring cardiologist DOLORES center.

ELIGIBILITY:
Inclusion Criteria:

* Patient who called UAS-ACS for a non-traumatic chest pain
* Patient who agreed to participate in the study.

Exclusion Criteria:

* Traumatic grief
* Patient refusal to participate in the observatory

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients that call to the SAMU-ACS because of chest pain
Sampling Method: Non-Probability Sample
Enrollment: 1816 (Actual)
Dates: Start 2009-11; Primary Completion 2011-11 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Direction | 1 day
  Matching the direction proposed by the ambulance and the final diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Christian Spaulding, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- French Society of Cardiology, Paris, France

REFERENCES:
- [Background] Bassand JP, Danchin N, Filippatos G, Gitt A, Hamm C, Silber S, Tubaro M, Weidinger F. Implementation of reperfusion therapy in acute myocardial infarction. A policy statement from the European Society of Cardiology. Eur Heart J. 2005 Dec;26(24):2733-41. doi: 10.1093/eurheartj/ehi673. Epub 2005 Nov 25. PMID 16311237
- [Background] Karlson BW, Herlitz J, Pettersson P, Ekvall HE, Hjalmarson A. Patients admitted to the emergency room with symptoms indicative of acute myocardial infarction. J Intern Med. 1991 Sep;230(3):251-8. doi: 10.1111/j.1365-2796.1991.tb00439.x. PMID 1895047
- [Background] Assez N, Adriansen C, Charpentier S, Baixas C, Ducasse JL, Goldstein P. [Management of acute coronary syndromes without ST elevation: the TOSCANE registry]. Arch Mal Coeur Vaiss. 2005 Nov;98(11):1123-9. French. PMID 16379109
- [Background] Bertrand ME, Simoons ML, Fox KA, Wallentin LC, Hamm CW, McFadden E, De Feyter PJ, Specchia G, Ruzyllo W; Task Force on the Management of Acute Coronary Syndromes of the European Society of Cardiology. Management of acute coronary syndromes in patients presenting without persistent ST-segment elevation. Eur Heart J. 2002 Dec;23(23):1809-40. doi: 10.1053/euhj.2002.3385. No abstract available. PMID 12503543
- [Background] Sauval P, Bout H, Ohanessian A, Danchin N, Monsegu J, Varenne O, Carli P, Spaulding C. [Management of chest pain by the Emergency Ambulance Service: the DOLORES register]. Arch Mal Coeur Vaiss. 2005 Nov;98(11):1095-9. French. PMID 16379105
- [Result] Manzo-Silberman S, Assez N, Vivien B, Tazarourte K, Mokni T, Bounes V, Greffet A, Bataille V, Mulak G, Goldstein P, Ducasse JL, Spaulding C, Charpentier S. Management of non-traumatic chest pain by the French Emergency Medical System: Insights from the DOLORES registry. Arch Cardiovasc Dis. 2015 Mar;108(3):181-8. doi: 10.1016/j.acvd.2014.11.002. Epub 2015 Feb 7. PMID 25662700